CLINICAL TRIAL: NCT06736353
Title: Effect of Classic Secondary Prevention in Type 2 MI: A Target Trial Emulation Study
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: TYPE2_MI_TARGET_TRIALS; KF10-0024 (Other Grant/Funding Number: The Swedish Foundation for Strategic Research)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Infarction Type 2
Keywords: Target trial emulation; Beta blocker; Statin; RAAS blocker; Single antiplatelet therapy; Dual antiplatelet therapy; Type 2 myocardial infarction; SWEDEHEART
MeSH Terms: interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Type 2 myocardial infarction: All patients reported as type 2 myocardial infarction (first reporting) in the Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART)
  Interventions: Drug: Beta Blocker Therapy or No Therapy (Control); Drug: RAAS blocker Therapy or No therapy (Control); Drug: Statin Therapy or No Therapy (Control); Drug: Single Antiplatelet Therapy or No Therapy (Control); Drug: Dual Antiplatelet Therapy or No Therapy (Control)

INTERVENTIONS:
Drug: Beta Blocker Therapy or No Therapy (Control) — Beta blocker therapy or no Beta blocker therapy initiated after type 2 myocardial infarction
Drug: RAAS blocker Therapy or No therapy (Control) — RAAS blocker therapy or no RAAS blocker therapy initiated after type 2 myocardial infarction
Drug: Statin Therapy or No Therapy (Control) — Statin therapy or no Statin therapy initiated after type 2 myocardial infarction
Drug: Single Antiplatelet Therapy or No Therapy (Control) — Single Antiplatelet Therapy or no antiplatelet therapy initiated after type 2 myocardial infarction
Drug: Dual Antiplatelet Therapy or No Therapy (Control) — Dual Antiplatelet Therapy or no Dual Antiplatelet Therapy initiated after type 2 myocardial infarction

SUMMARY:
A classic heart attack is caused by a blockage to the coronary arteries that supplies the heart muscle with oxygenated blood. The medical term for this condition is type 1 myocardial infarction. There is strong scientific evidence that the usage of pharmacological drugs such as statins, beta blockers, Renin-Angiotensin-Aldosterone System blockers and platelet inhibitors after a type 1 myocardial infarction improves survival and reduces the risk for new myocardial infarctions. However, a myocardial infarction may also occur without blockage to the coronary arteries when other acute conditions causes either a decreased supply or an increased demand of oxygenated blood to the heart. The medical term for the latter is type 2 myocardial infarction. There are currently no scientific evidence that any pharmacological drug improves survival in patients with a type 2 myocardial infarction, of whom only one in three patients are alive after five years.

The aim of this study is to investigate if those drugs that improves the prognosis after a type 1 myocardial infarction (Beta blockers, Renin-Angiotensin-Aldosterone System blockers, Statins and platelet inhibitors) also affects the prognosis after a type 2 myocardial infarction.

The best way to answer this question would be to conduct clinical trials for each drug where type 2 myocardial infarction patients are randomized to either receiving the drug of interest or receiving placebo (sugar pills) and then compare the survival and outcomes in both groups over time.

However, clinical trials are costly, time consuming and also difficult to conduct with type 2 myocardial infarction patients since these patients are treated at various hospital departments.

Therefore, this study will instead include patients in a Swedish national register for myocardial infarction, in which myocardial infarction patients are reported from all Swedish hospitals, and compare type 2 myocardial infarction patients that did receive or did not receive each treatment. To minimize the risk of making inaccurate conclusions about the causal relationship between treatment and outcome, the study will define the optimal clinical trial for each treatment and then specifically emulate these trials in all possible aspects using the register data. This method is called "target trial emulation".

DETAILED DESCRIPTION:
While acute and long term treatments in type 1 myocardial infarction (MI) are well documented, there are no evidence based treatments altering the prognosis in type 2 MI patients, of whom only one in three are alive after five years. Classic secondary preventive treatment in type 1 MI include the use of statins, beta blockers, renin-angiotensin-aldosterone system (RAAS) inhibitors, single antiplatelet therapy (SAPT) and dual antiplatelet therapy (DAPT). While some observational studies suggest classic secondary preventive MI treatment to be associated with better survival in type 2 MI, others do not.

The aim of this study is to investigate if there is an association between treatment with each of statins, beta blockers, RAAS inhibitors, SAPT or DAPT; and all-cause mortality or long-term cardiovascular events in patients with type 2 MI.

The study will be conducted as (several) registry-based observational studies emulating pre-specified target trials. A protocol of a pragmatic randomized controlled trial (a target trial) will be specified for each of statins, beta blockers, RAAS inhibitors, SAPT and DAPT; including eligibility criteria, treatment assignment, time zero and follow up, outcomes, causal contrast and statistical analyses.

Each of these components will then be emulated using registry data. The target trial, as well as the registry-based study emulating the target trial, will differ slightly for each treatment.

The study will include all, approximately 14 000, patients reported as type 2 MI (first reporting for each patient) in the Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART) from 2010 and onward. Data from SWEDEHEART will be merged with data from the National Patient Register, the Swedish Cause of Death Register and the Longitudinal Integrated Database for Health Insurance and Labour Market Studies.

Patients will be followed from hospital discharge (time zero) until death, loss to follow-up or end of follow up (date of data collection). Treatment specific eligibility criteria will be applied at time zero. All important confounding factors at time zero will be identified by drawing causal diagrams, one for each treatment and outcome. Treatment specific models with registry data will then be created to balance the assigned groups using for example inverse probability weighting with multiple imputation of missing data among covariates.

For all target trial emulations, the primary outcome of interest will be a composite endpoint of all-cause mortality, readmission for MI, stroke or heart failure. Secondary outcomes will be all-cause mortality, cardiovascular mortality, readmission for MI, readmission for stroke and readmission for heart failure individually. Safety outcomes will be specified separately for each treatment. Readmission for bacterial pneumonia will be used as a negative control outcome in all target trial emulations to check for residual confounding. Intention-to-treat analysis will be performed for each treatment and outcome. Competing risk methodology will be applied as appropriate.

ELIGIBILITY:
Beta blocker target trial emulation:

Inclusion Criteria:

* Reported as Type 2 MI in SWEDEHEART
* Age >18 years
* Alive at time zero (hospital discharge)

Exclusion Criteria:

* Already on beta blocker
* Heart failure with reduced ejection fraction
* Hypertrophic obstructive cardiomyopathy
* Systolic blood pressure <90 mmHg
* Heart rate <50 bpm
* Metastatic cancer (proxy for terminal disease)
* History of dementia or substance abuse last 6 months (proxy for unable to adhere to treatment)
* Missing data for any exclusion criteria

RAAS blocker target trial emulation:

Inclusion Criteria:

* Reported as Type 2 MI in SWEDEHEART
* Age >18 years
* Alive at time zero (hospital discharge)

Exclusion Criteria:

* Already on RAAS blocker
* Heart failure with reduced ejection fraction
* Combination of prior myocardial infarction and diabetes mellitus
* Diabetic nephropathy,
* Systolic blood pressure <90 mmHg
* Hyperkalemia
* Acute renal failure
* Pregnancy
* Metastatic cancer (proxy for terminal disease)
* History of dementia or substance abuse last 6 months (proxy for unable to adhere to treatment)
* Missing data for any exclusion criteria

Statin target trial emulation:

Inclusion Criteria:

* Reported as Type 2 MI in SWEDEHEART
* Age >18 years
* Alive at time zero (hospital discharge)

Exclusion Criteria:

* Already on Statin
* Revascularization during hospitalization
* Obstructive coronary artery disease detected during hospitalization
* History of myocardial infarction or coronary revascularization
* History of stroke
* History of peripheral artery disease
* Familial hypercholesterolemia
* Pregnancy
* Acute or chronic liver failure
* Metastatic cancer (proxy for terminal disease)
* History of dementia or substance abuse last 6 months (proxy for unable to adhere to treatment)
* Missing data for any exclusion criteria

Single Antiplatelet Therapy target trial emulation:

Inclusion Criteria:

* Reported as Type 2 MI in SWEDEHEART
* Age >18 years
* Alive at time zero (hospital discharge)

Exclusion Criteria:

* Already on antiplatelet therapy
* Revascularization during hospitalization
* Obstructive coronary artery disease detected during hospitalization
* Indication for dual antiplatelet therapy according to treating physician
* History of myocardial infarction or coronary revascularization
* History of stroke
* History of peripheral artery disease
* Severe anemia (Hemoglobin <90g/L)
* Intracranial or gastrointestinal bleeding within the last 12 months
* Bleeding disorder
* Acute bleeding during hospitalization
* Metastatic cancer (proxy for terminal disease)
* History of dementia or substance abuse last 6 months (proxy for unable to adhere to treatment)
* Missing data for any exclusion criteria

Dual Antiplatelet Therapy target trial emulation:

Inclusion Criteria:

* Reported as Type 2 MI in SWEDEHEART
* Age >18 years
* Alive at time zero (hospital discharge)

Exclusion Criteria:

* Already on Dual Antiplatelet Therapy
* Revascularization during hospitalization
* Severe anemia (Hemoglobin <90g/L)
* Pregnancy
* Treatment with oral anticoagulants
* Intracranial or gastrointestinal bleeding within the last 12 months
* Bleeding disorder
* Acute bleeding during hospitalization
* Metastatic cancer (proxy for terminal disease)
* History of dementia or substance abuse last 6 months (proxy for unable to adhere to treatment)
* Missing data for any exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients reported as type 2 myocardial infarction (first reporting) in the Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART). SWEDEHEART is a Swedish national register for coronary artery disease care and valvular interventions. All Swedish hospitals report to SWEDEHEART. Reported myocardial infarction patients have been classified into type 1-5 since 2010 by the reporting physician. All patients will be included, from the first reporting, until the date of data collection.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2010-09-03 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Composite | From enrollment (hospital discharge after type 2 MI) until Composite endpoint, Loss to follow-up or End of follow up (date of data collection: 05-May-2022)
  Composite endpoint: All-cause mortality, readmission for MI, stroke or heart failure

SECONDARY OUTCOMES:
All-cause mortality | From enrollment (hospital discharge after type 2 MI) until Death, Loss to follow-up or End of follow up (date of data collection: 05-May-2022)
  Death from any cause
Cardiovascular mortality | From enrollment (hospital discharge after type 2 MI) until Cardiovascular death, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Death from cardiovascular disease
Readmission for MI | From enrollment (hospital discharge after type 2 MI) until Readmission for MI, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Readmission for myocardial infarction
Readmission for stroke | From enrollment (hospital discharge after type 2 MI) until Readmission for Stroke, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Readmission for stroke
Readmission for heart failure | From enrollment (hospital discharge after type 2 MI) until Readmission for Heart failure, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Readmission for heart failure

OTHER OUTCOMES:
Readmission for Asthma or COPD | From enrollment (hospital discharge after type 2 MI) until Readmission for Asthma/COPD, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Safety outcome in Beta blocker target trial emulation. Readmission for Asthma or Chronic Obstructive Pulmonary Disease. Only if main diagnosis.
Readmission for Acute renal failure | From enrollment (hospital discharge after type 2 MI) until Readmission for Acute renal failure, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Safety outcome in RAAS blocker target trial emulation. Readmission for Acute renal failure.
Readmission for bleeding | From enrollment (hospital discharge after type 2 MI) until Readmission for Bleeding, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Safety outcome in SAPT and DAPT target trial emulations. Readmission for bleeding.
Readmission for Pneumonia | From enrollment (hospital discharge after type 2 MI) until Readmission for bacterial pneumonia, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Negative control outcome in all target trial emulations. Readmission for bacterial pneumonia.
Readmission for hip fracture | From enrollment (hospital discharge after type 2 MI) until Readmission for hip fracture, Loss to follow-up or End of follow up (date of data collection: 05-May-2022). Competing risk methodology applied.
  Additional negative control outcome in all target trial emulations. Readmission for hip fracture.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of medical sciences, Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Due to Swedish laws on personal integrity and health data, as well as the Ethics Committee, we are not allowed to make any data included health variables open to the public even if made anonymous. The data could be shared with other researchers after a request to the head of our department